CLINICAL TRIAL: NCT03058679
Title: Open Label, Randomized, Multicenter, Comparative Effectiveness Trial of Specific Carbohydrate and Mediterranean Diets to Induce Remission in Patients With Crohn's Disease
Brief Title: Trial of Specific Carbohydrate and Mediterranean Diets to Induce Remission of Crohn's Disease
Acronym: DINE-CD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Crohn's and Colitis Foundation (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 825907
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Results first posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-06

CONDITIONS: Crohn Disease
Keywords: diet; specific carbohydrate diet; Mediterranean style diet; randomized controlled trial
MeSH Terms: conditions — Crohn Disease | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Specific Carbohydrate Diet (Experimental): For the first six 6 weeks of the trial, participants received a weekly delivery of prepared meals compliant with the SCD (breakfast, lunch, dinner, and two 2 snacks per day). Meals were prepared by Healthy Chef Creations (Orlando, FL) based on menus developed by the food vendor in consultation with study dietitians. Participants assigned to the SCD received a three3-day starter diet as recommended in Breaking the Vicious Cycle. Meals were designed to be heated in an oven or microwave. No other preparation was required.
  Interventions: Other: Diet
- Mediterranean Style Diet (Active Comparator): For the first six 6 weeks of the trial, participants received a weekly delivery of prepared meals compliant with the MD (breakfast, lunch, dinner, and two 2 snacks per day). Meals were prepared by Healthy Chef Creations (Orlando, FL) based on menus developed by the food vendor in consultation with study dietitians. Meals were designed to be heated in an oven or microwave. No other preparation was required.
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — food for the diet will be provided to the participants for 6 weeks and participants will follow the diet on their own for the remaining 6 weeks

SUMMARY:
This protocol is designed to compare the effectiveness of two dietary interventions for patients with Crohn's disease (CD): the Specific Carbohydrate Diet (SCD) and a Mediterranean style diet (MSD) that has been demonstrated to have numerous other health benefits. The two diets will be compared in terms of their ability to resolve both the symptoms and bowel inflammation that characterize this debilitating disease.

DETAILED DESCRIPTION:
This study tested whether the SCD is superior to a MSD for managing symptoms and reducing inflammatory markers in patients with CD.

The study was designed to include 194 patients with CD who have 1) active symptoms defined by a short Crohn's Disease Activity Index (sCDAI) score >175. Although the initial plan was to also require that all patients have active inflammation documented by a fecal calprotectin (FCP) concentration >250mcg/g or high sensitivity C-reactive protein (CRP) >7 mg/L or ulceration of the small bowel and/or colon consistent with an SES-CD score >4 as documented in routine clinical practice within 4 weeks of screening, a decision was made early in the recruitment period to enroll all patients with CD with sCDAI>175 regardless of the results of the tests for inflammatory markers and to perform subgroup analyses of those with and without evidence of inflammation.

Eligible participants were randomly assigned to follow one of the diets in a 1:1 ratio. Participants were provided with 3 meals and 2 snacks each day for a period of 6 weeks. The meals and snacks were prepared by the food vendor, Healthy Chef Creations, and were delivered directly to the participant's home once per week. Participants in both groups were also provided with instructions on how to follow the diets on their own. Participants reported their symptoms through an electronic diary and provided stool samples for FCP measurement and blood for CRP measurement at weeks 0, 6 and 12. The primary and secondary outcomes were assessed at week 6. Following week 6, participants were able to pay out of pocket to purchase food from Healthy Chef Creations and/or could attempt to follow their assigned diet completely on their own. At week 12, in addition to the primary and secondary outcomes assessed again

ELIGIBILITY:
Inclusion Criteria

1. Age ≥18
2. Documented diagnosis of Crohn's disease
3. sCDAI score >175
4. Documentation of receipt of a baseline stool sample by the data coordinating center and hsCRP.
5. Access to a computer with internet and the ability to complete daily online surveys
6. Capable of providing consent to participate
7. Able to receive weekly food shipments delivered every Friday for 6 weeks

Exclusion Criteria

1. Pregnancy
2. sCDAI >400
3. Hospitalized patients
4. Anticipated need for surgery within 6 weeks of randomization
5. Use of the Specific Carbohydrate Diet within 4 weeks of screening
6. Start or change*** dose of thiopurines (azathioprine and 6-MP), methotrexate, natalizumab, or vedolizumab within 12 weeks prior to screening
7. Start or change*** dose of anti-tumor necrosis factor (TNF) agents (including infliximab (Remicade), adalimumab (Humira), certolizumab pegol (Cimzia), golimumab (Simponi) or ustekinumab within 8 weeks prior to screening.
8. Start or change in dose of any 5-aminosalicylic acid (5-ASA) medications within 2 weeks of screening.
9. Start or change dose of corticosteroids within 1 week of screening or a dose >20mg/day prednisone or equivalent*
10. Use of antibiotics (other than topical formulations) for any reason within 2 weeks prior to screening
11. Known symptomatic intestinal stricture.
12. Presence of an ostomy
13. Baseline stool frequency >4 bowel movements/day when well
14. BMI <16
15. BMI ≥40
16. Celiac disease
17. Documented C difficile colitis within four weeks of screening
18. Diabetes Mellitus requiring medication
19. Albumin<2.0mg/dl, within 4 weeks of screening (if tested as part of routine clinical care)
20. Known allergy to tree nuts or peanuts
21. Other conditions that would be a contraindication to any of the study diets or preclude the participant from completing the study.
22. Currently participating in another clinical trial of a drug to treat Inflammatory Bowel Disease (IBD) or a dietary therapy for any indication.

    * Patients may continue these medications at stable dose for the first six weeks and budesonide may be used at any dose. After the 6th week in the study, patients may taper their steroid dose. The study will provide a recommended taper schedule.

      * Loading/induction doses of biologic type medication will be considered a stable doses. ***Exception for treatment failures: if a subject is determined to fail on any of the following standard lines of treatment at the treating investigator's discretion, subjects may screen for study intervention based upon the following wash out periods: 4 weeks for thiopurine and methotrexate and 8 weeks for natalizumab, vedolizumab, anti-TNF, or ustekinumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D Lewis, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (35):
- United States (35):
  - University of Arizona, Tucson, Arizona
  - UCSF Colitis and Crohn's Disease Center, San Francisco, California
  - University of Colorado Denver, Denver, Colorado
  - Emory University, Atlanta, Georgia
  - Atlanta Gastroenterology, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - Northwestern University, Evanston, Illinois
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - The University of Louisville, Louisville, Kentucky
  - University of Maryland Baltimore, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Clinical Research Institute of Michigan, Chesterfield, Michigan
  - Troy Gastroenterology, Troy, Michigan
  - The University of Minnesota, Minneapolis, Minnesota
  - Minnesota Gastroenterology, P.A, Plymouth, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - NYU Langone Medical Center, New York, New York
  - Weill Cornell - NewYork Presbyterian, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Lenox Hill Hospital, New York, New York
  - The University of North Carolina, Chapel Hill, North Carolina
  - Atrium Health (formerly Carolinas HealthCare System), Charlotte, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio State University - Wexner Medical Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Lifespan Health System, Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lewis JD, Sandler RS, Brotherton C, Brensinger C, Li H, Kappelman MD, Daniel SG, Bittinger K, Albenberg L, Valentine JF, Hanson JS, Suskind DL, Meyer A, Compher CW, Bewtra M, Saxena A, Dobes A, Cohen BL, Flynn AD, Fischer M, Saha S, Swaminath A, Yacyshyn B, Scherl E, Horst S, Curtis JR, Braly K, Nessel L, McCauley M, McKeever L, Herfarth H; DINE-CD Study Group. A Randomized Trial Comparing the Specific Carbohydrate Diet to a Mediterranean Diet in Adults With Crohn's Disease. Gastroenterology. 2021 Sep;161(3):837-852.e9. doi: 10.1053/j.gastro.2021.05.047. Epub 2021 May 27. PMID 34052278

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 33 clinical sites across the United States. Enrollment in the trial occurred between September 29, 2017 and October 8, 2019.
Pre-assignment Details: There were 3 main reasons that participants who consented to the study were not randomized. The majority did not meet eligibility criteria. A small number withdrew or were lost to follow-up
Groups:
- Specific Carbohydrate Diet; Mediterranean Style Diet: Diet: food for the diet will be provided to the participants for 6 weeks
Period: Baseline to Week 6
Arm/Group | Specific Carbohydrate Diet | Mediterranean Style Diet
Started | 99 (3 randomized to SCD withdrew before starting diet;2 randomized pts w/ baseline sCDAI<150 excluded.) | 92 (Due to an error 1 participant was randomized with a baseline sCDAI<150. This pt was excluded.)
Completed | 81 | 77
Not Completed | 18 | 15
Not completed — Lost to Follow-up | 3 | 2
Not completed — Change in Crohn's disease medication | 4 | 2
Not completed — Adverse Event | 6 | 6
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Difficulty following the diet | 0 | 2
Not completed — Physician Decision | 1 | 0
Period: Week 6 to Week 12
Arm/Group | Specific Carbohydrate Diet | Mediterranean Style Diet
Started | 81 | 77
Completed | 61 | 60
Not Completed | 20 | 17
Not completed — Change in medication | 5 | 7
Not completed — Adverse Event | 4 | 3
Not completed — Withdrawal by Subject | 9 | 4
Not completed — Difficulty following the assigned diet | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mediterranean Style Diet | Specific Carbohydrate Diet | Total
Number analyzed (Participants) | 92 | 99 | 191
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 37.0 [29.5 to 53.0] | 36.0 [27.0 to 46.0] | 37 [28.0 to 50.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 58 | 121
  Male | 29 | 41 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 88 | 92 | 180
  Unknown or Not Reported | 0 | 3 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 2 | 2
  Black | 2 | 5 | 7
  Multiracial | 1 | 1 | 2
  Other | 3 | 1 | 4
  Unknown | 0 | 2 | 2
  White | 86 | 88 | 174
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m2] | 25.1 [21.3 to 29.9] | 25.6 [22.5 to 29.0] | 25.3 [21.8 to 29.5]
Smoking status [Count of Participants; unit: Participants]
  Never | 68 | 79 | 147
  Past | 21 | 20 | 41
  Current | 3 | 0 | 3
Years since CD diagnosis [Median (Inter-Quartile Range); unit: years] | 10 [5 to 21] | 10 [3 to 16] | 10 [4 to 17]
CD behavior [Count of Participants; unit: Participants]
  Non-stricturing, nonpenetrating | 56 | 60 | 116
  Stricturing | 19 | 17 | 36
  Penetrating | 9 | 13 | 22
  Stricturing and penetrating | 8 | 9 | 17
Crohn's disease distribution [Count of Participants; unit: Participants]
  Ileum alone | 22 | 30 | 52
  Colon alone | 17 | 13 | 30
  Ileum and Colon | 53 | 55 | 108
  Missing | 0 | 1 | 1
History of perianal fistula [Count of Participants; unit: Participants] | 24 | 20 | 44
History of intestinal surgery [Count of Participants; unit: Participants] | 34 | 29 | 63
Current use of any biologic [Count of Participants; unit: Participants] | 55 | 53 | 108
Current use of immunomodulators [Count of Participants; unit: Participants] | 11 | 11 | 22
Current use of oral 5-ASA [Count of Participants; unit: Participants] | 6 | 15 | 21
Current use of rectal 5 ASA [Count of Participants; unit: Participants] | 0 | 3 | 3
Current use of oral steroids [Count of Participants; unit: Participants] | 3 | 11 | 14
Current use of rectal steroids [Count of Participants; unit: Participants] | 1 | 2 | 3
Number of prior anti-TNF medications [Count of Participants; unit: Participants]
  0 | 28 | 34 | 62
  1 | 22 | 29 | 51
  2 | 32 | 26 | 58
  3 | 9 | 9 | 18
  4 | 1 | 1 | 2
Prior ustekinumab [Count of Participants; unit: Participants] | 22 | 23 | 45
Prior vedolizumab [Count of Participants; unit: Participants] | 27 | 22 | 49
hsCRP mg/L [Median (Inter-Quartile Range); unit: mg/L] | 2.5 [1.2 to 6.2] | 3.2 [1.4 to 8.1] | 2.9 [1.4 to 7.5]
hsCRP >5 mg/L [Count of Participants; unit: Participants] | 28 | 37 | 65
fecal calprotectin (FC) ug/g [Median (Inter-Quartile Range); unit: ug/g] | 40.0 [16.0 to 185.0] | 107.5 [16.0 to 223.0] | 70 [16.0 to 194.0]
fecal calprotectin (FC) >250 ug/g [Count of Participants; unit: Participants] | 13 | 23 | 36
Inflammation on colonoscopy [Count of Participants; unit: Participants]
  Not performed | 80 | 89 | 169
  Yes | 8 | 8 | 16
  Probably | 1 | 0 | 1
  Probably not | 1 | 1 | 2
  No | 2 | 1 | 3
FC>250 ug/g or hsCRP>5 mg/L or definite inflammation on colonoscopy [Count of Participants; unit: Participants] | 38 | 50 | 88
sCDAI (median, Q1-Q3) [Median (Inter-Quartile Range); unit: units on a scale] — Short Crohn's Disease Activity Index. This is a method to measure Crohn's disease patient's symptoms using only a questionnaire,which can be completed without an office visit or lab work. The variables included in the short CDAI are abdominal pain, diarrhea frequency, and general well-being. The higher the score, the worse the disease activity. The sCDAI uses the same scale as the full CDAI, such that scores,<150 define remission, 150 to 219 mild activity, 220 to450 moderate activity, and.450 severe activity. The total score is reported.
  units on a scale | 217.7 [195.7 to 247.0] | 226.0 [197.0 to 263.8] | 223.0 [195.7 to 259.6]
CDAI (median, Q1-Q3) [Median (Inter-Quartile Range); unit: units on a scale] — The Crohn's Disease Activity Index - CDAI scores range from 0 to 600. A score of less than 150 denotes relative disease quiescence (remission); 150 to 219, mildly active disease; 220 to 450, moderately active disease; and greater than 450, severe disease. The higher the score, the worse the disease activity.
  This index uses the following variables to determine a score: number of stools, abdominal pain, general well-being, extraintestinal complications, antidiarrheal agents used in the previous 7 days, abdominal mass felt on palpation, hematocrit, and body weight
  units on a scale | 206.8 [179.3 to 247.0] | 210.0 [169.8 to 246.2] | 209.5 [171.5 to 246.2]
Short IBDQ (median, Q1-Q3) [Median (Inter-Quartile Range); unit: units on a scale] — The SIBDQ is a 10-item health-related quality of life (HRQOL) questionnaire validated for use in CD patients. It assesses physical, social, and emotional status and is scored on a 7-point Likert scale from 1 (severe problem) to 7 (no problems at all). Scores for each question are summed to provide a total score. The total score is reported. The absolute score ranges from 10 (poor HRQOL) to 70 (optimum HRQOL).
  units on a scale | 38.0 [33.0 to 44.0] | 40.0 [33.0 to 45.0] | 39.0 [33.0 to 45.0]
PROMIS measures (median, Q1-Q3) [Median (Inter-Quartile Range); unit: units on a scale] — Patient-Reported Outcomes Measurement Information System (PROMIS)- set of person-centered measures that evaluate and monitor health status. All assessments are for the last 7 days. To calculate a total raw score, each item is scored on a scale of 1-5. If the form has 7 items, the lowest possible raw score is 7 and the highest possible raw score is 35. Raw scores are then translated into T scores. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. T-scores are reported. Higher T-scores denote worse outcomes.
  units on a scale
    Fatigue | 60.4 [55.9 to 65.9] | 58.9 [54.8 to 65.6] | 59.6 [55.0 to 65.8]
    Pain interference | 60.1 [55.7 to 63.8] | 61.3 [55.7 to 63.6] | 61.2 [55.7 to 63.7]
    Sleep disturbance | 57.3 [51.4 to 62.1] | 54.5 [49.4 to 60.2] | 56.0 [50.9 to 61.4]
    Social isolation | 48.4 [41.0 to 56.1] | 47.2 [34.8 to 53.8] | 47.9 [34.8 to 54.5]
Inflammatory back pain screen [Count of Participants; unit: Participants] — This self-reported survey assessed five criteria defining possible inflammatory back pain:(1) improvement with exercise (2) pain at night (3) insidious onset (4) age at onset <40 years and (5) no improvement with rest. The higher the score the more likely the person had inflammatory back pain.
  Participants
    0 | 30 | 40 | 70
    1-3 | 39 | 40 | 79
    >3 | 22 | 18 | 40
    Missing | 1 | 1 | 2
AMeD Score [Median (Inter-Quartile Range); unit: units on a scale] — Alternate Mediterranean Diet Score - Participants completed a 24-hour dietary recall at baseline, during week 6 and during week 12. These data were used to compute the Alternate Mediterranean Diet Score (AMeD) where a higher score implies greater consistency with a Mediterranean diet. AMeD scores range from 0 (minimal adherence) to 9 (maximal adherence).
  units on a scale | 3.0 [1.0 to 4.0] | 2.0 [1.0 to 3.0] | 3.0 [2.0 to 4.0]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants That Achieved Symptomatic Remission at Week 6
Description: Assessed by Short Crohn's Disease Activity Index (sCDAI) - diarrhea, abdominal pain and general well being; sCDAI <150 in the absence of initiation or increase of any CD medications
Time Frame: 6 weeks
Population: percentage of participants who achieved symptomatic remission at week 6
Measure: Count of Participants; unit: Participants
Arm/Group | Mediterranean Style Diet | Specific Carbohydrate Diet
Number analyzed (Participants) | 92 | 99
Participants | 40 | 46

2. Primary Outcome: Reduction in Bowel Inflammation Among Those Whose Screening Fecal Calprotectin (FC) Was Greater Than 250μg/g at Baseline and Who Had an FC Results at Both Baseline and Week 6
Description: reduction of calprotectin to less than 250 μg/g and by greater than 50% from screening among those with screening FC >250 μg/g
Time Frame: 6 weeks
Population: This measure includes only those whose screening fecal calprotectin (FC) was greater than 250μg/g at baseline and who had an FC results at both baseline and week 6
Measure: Count of Participants; unit: Participants
Arm/Group | Mediterranean Style Diet | Specific Carbohydrate Diet
Number analyzed (Participants) | 13 | 23
Participants | 4 | 8

3. Secondary Outcome: Percentage of Participants That Reached Clinical Remission at Week 6
Description: Assessed by the CDAI - CDAI <150
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mediterranean Style Diet | Specific Carbohydrate Diet
Number analyzed (Participants) | 92 | 99
Participants | 44 | 48

4. Secondary Outcome: Percentage of Participants With a Reduction in Systemic Inflammation at Week 6
Description: reduction in high-sensitivity CRP (hsCRP) to <5 mg/L and >50% reduction from screening among those with screening hsCRP >5mg/L
Time Frame: 6 weeks
Population: This measure includes only those that had a screening hsCRP > 5mg/L and had hsCRP measured at both screening and at week 6
Measure: Count of Participants; unit: Participants
Arm/Group | Mediterranean Style Diet | Specific Carbohydrate Diet
Number analyzed (Participants) | 28 | 37
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: AEs were recorded at each study contact from screening visit to a participant's end of study visit. For participants that completed the study, AEs were assessed at screening, baseline, wk 6 and week 12. Among participants who withdrew early from the study, AEs were assessed at the above named timepoints until the time of withdraw. The clinical course of each AE was followed until resolution, stabilization, or until it was determined that study intervention or participation was not the cause.
Description: As per the DINE-CD protocol, allergic reaction to a component of the food, intolerance of the food other than allergic reaction, worsening of CD and worsening of extraintestinal manifestations of CD was considered expected. AEs were included for all randomized participants who started the diet with the exception of 3 participant who were randomized in error with an sCDAI <150 (as noted in the participant flow).
Arm/Group | Mediterranean Style Diet | Specific Carbohydrate Diet
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/99
Serious Adverse Events (participants affected / at risk) | 5/92 | 3/99
Other Adverse Events (participants affected / at risk) | 18/92 | 19/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mediterranean Style Diet (N=92) | Specific Carbohydrate Diet (N=99)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (3)
Worsening of Crohn's disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mediterranean Style Diet (N=92) | Specific Carbohydrate Diet (N=99)
Abdominal pain (Gastrointestinal disorders) | 13 (14) | 10 (11)
Diarrhea (Gastrointestinal disorders) | 7 (7) | 5 (5)
Gastrointestingal disorders other - Worsening of Crohn's disease symptons (Gastrointestinal disorders) | 4 (4) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/79/NCT03058679/Prot_SAP_000.pdf